CLINICAL TRIAL: NCT06719076
Title: IMPACT OF DIABETES HEALTHCARE PROGRAM ON GLYCEMIC CONTROL AND SELF-EFFICACY AMONG TYPE-II DIABETICS IN ISLAMABAD PAKISTAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Services Academy, Islamabad, Pakistan (Other)
Responsible Party: Principal Investigator, Abdul Samad, Principle Investigator, Health Services Academy, Islamabad, Pakistan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000574/HSA/MSPH-2023
Record Dates: First submitted 2024-11-26; First posted 2024-12-05 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: HbA1c
Keywords: HBA1c levels; RCT Pakistan; Self-Efficacy; T2DM; Diabetes Mellitus; Glucose Metabolism Disorders
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders

STUDY DESIGN:
Intervention Model Description: In single group arm design the Type-II Diabetics randomized in two arms the first arm receive 3 months of DHCP intervention and other arm receive 3 month usual care. The allocation of groups assigned after the randomization either for intervention arm or control arm and the result will be compared and interpreted and disseminated.
Masking Description: To maintain internal validity and minimize bias, randomization will be employed to allocate participants to either the control group or the Diabetes Healthcare Program group. A series of individually concealed envelopes will be prepared by an assistant not involved in the trial (Clark et al., 2021). Each bearing a randomly assigned indication of either "Control group" or "Diabetes Healthcare Program group" and sequentially numbered. Once a participant provides informed consent and meets the inclusion criteria, the next envelope in line will be opened to determine the group allocation, ensuring that randomization remains blinded to the research team until allocation is revealed. This approach adheres to the CONSORT guidelines, which recommend randomization in trials to avoid confounding variables and ensure comparability between groups (Schulz et al., 2010).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diabetes Healthcare Program DHCP (Experimental): Type-II Diabetics in the intervention group will be received for 3 months of DHCP as well as usual care. Additional for session participation reminders messages will be sent 3 days before training and the messages will be forwarded by Principal Investigator and Research Assistant. Outcome variable will be measured at two points at the baseline and after completing of 3 months of intervention.
  Interventions: Behavioral: Diabetes Healthcare Program (DHCP)
- No intervention arm (No Intervention): Type-II Diabetes in the control group will receive usual care, which includes routine consultations with physicians and pharmacological therapy as prescribed by healthcare provider. The frequency of clinic visits will be every 3 months, with monitoring of blood glucose levels, blood pressure, and lipid profiles. The usual care protocol is based on the guidelines for the management of type 2 diabetes mellitus by the American Diabetes Association (Care, 2023)

INTERVENTIONS:
Behavioral: Diabetes Healthcare Program (DHCP) — Training for Type-II Diabetics
  The program includes 6 structured training sessions, each session will delivered biweekly and lasting for 1 hour and 20 minutes , covering topics such as:
  Week 1: Diabetes Education and Goal Setting Week 3: Nutrition and Meal Planning Week 5: Physical Activity and Exercise Week 7: Medication Management Week 9: Stress Management and Emotional Well-being Week 11: Review and Future Plans Time, Venue, and Interactive Activities Sessions will be held at the Federal General Hospital Basement, on Fridays, from 10:00 am to 11:20 am. Each session includes interactive elements, such as group discussions, practical exercises, and hands-on activities, to ensure participants are fully engaged and equipped to manage their T2DM diabetes.
  Arms: Diabetes Healthcare Program DHCP

SUMMARY:
Type 2 Diabetes Mellitus (T2DM) is a significant public health challenge in Pakistan, characterized by a growing prevalence and substantial economic burden. The alarming rise in T2DM cases in Pakistan highlights the need for evidence-based solutions to control the disease. However, there is a notable knowledge gap in the effectiveness of diabetes healthcare program interventions in Pakistan.

The goal of this randomized controlled trial (RCT) is to evaluate the effectiveness of a Diabetes Healthcare Program in improving glycemic control and enhancing Self-efficacy in Type-II Diabetic patients in Islamabad, Pakistan. The main questions it aims to answer are whether the Diabetes Healthcare Program can reduce HbA1c levels and enhance Self-efficacy in Type-II Diabetic patients. Researchers will compare the outcomes of 37 patients receiving the Diabetes Healthcare Program with 37 patients receiving standard care to see if the program improves glycemic control and enhances Self-efficacy. Participants will attend 12 weeks of Diabetes Healthcare Program sessions, receive standard care from the hospital's diabetes department, and complete surveys and questionnaires to assess their Self-efficacy and glycemic control at baseline and after the 3 months intervention period.

DETAILED DESCRIPTION:
Objective: To evaluate the impact of Diabetes Healthcare Program on reducing HbA1c levels and enhance Self-efficacy in Type-II Diabetics in Islamabad.

Setting, Duration, Study Type: The study was carried out as a randomized controlled trial (RCT) in Federal General Hospital Islamabad, which will be completed in 6 months. The study protocols was approved by ethical review board of Health Services Academy under letter no 000574/HSA/MSPH-2023 dated 23- Aug-2024. throughout the recruitment process.

Methods: A total of 74 Type-II Diabetics were invited to participate in the study, and those who visited the hospital underwent the recruitment process using a concealed envelop method. Recruitment was stopped once the required sample size of 74 participants was met. Using random allocation, 37 subjects were assigned to the control group and 37 to the intervention group. Both the control group and the intervention group received usual care delivered at FGH. The intervention group additionally received a Diabetes Health Care Program Intervention for 12-week duration.

Expected Outcome: The study aims to demonstrate that the Diabetes Healthcare Program (DHCP) intervention group will have enhanced Self-efficacy scores and reduced HbA1c levels compared to the control group among Type-II Diabetics in Islamabad. If successful, the study's findings will be generalizable to similar settings worldwide, contributing significantly to the existing body of literature on improving glycemic control and Self-efficacy in Type-II Diabetes. The study's results will have practical implications, informing policymakers on the development of evidence-based strategies to manage type II diabetes at a national level. This will ultimately enable the creation of targeted interventions and policies to improve the health outcomes of individuals with type II diabetes, contributing to global efforts to combat this growing health concern.

ELIGIBILITY:
Inclusion Criteria:

* Type-II Diabetes on follow-up treatment in FGH for last 6 months.
* Type-II Diabetic age 18 years and above of both genders.
* Type-II Diabetic with uncontrolled Diabetes whose HbA1c reading is >7% at last assessment within 3 months
* Type-II Diabetic living in Islamabad.

Exclusion Criteria:

* Type-II Diabetic recognized as disabled and suffering from loss of hearing.
* Type-II Diabetics with serious complications such as retinopathy/kidney disease/tachycardia in a stable status > 100/minute, or serious diabetic feet
* Type-II Diabetic currently using injection insulin impaired glucose tolerance, metabolic syndrome, maturity onset diabetes of youth and gestational diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-01-26 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Glycemic Control (HbA1c Levels) | The primary outcome will be measured at two time points: first at baseline and second after 3 months following the implementation of the intervention.
  The HbA1c test is a widely used indicator of glycemic control, reflecting the average blood glucose concentration over the preceding 2-3 months. The level of HbA1c is influenced by the blood glucose concentration, the duration of red blood cell exposure to varying concentrations, and the quantity of red blood cells. The HbA1c test has been reviewed and validated in numerous studies (Sherwani et al., 2016). The score ranges from 5% to 15%, with a normal score of 5.7% or less, a prediabetes score of 5.8% to 6.4%, and a diabetes score of 6.5% or higher.

SECONDARY OUTCOMES:
Enhance Self-efficacy | The secondary outcome will be measured at two time points: first at baseline and second after 3 months following the implementation of the intervention.
  Self-efficacy is a crucial component of Social Cognitive Theory in diabetes management. The Diabetes Management Self-efficacy Scale (DMSES) will be used to assess Self-efficacy in diabetes management. The DMSES measures confidence in conducting self-care activities, such as blood sugar monitoring, healthy eating, and physical activity. The scale ranges from 0 to 200, categorizing Self-efficacy into low (0-79), moderate (80-119), high (120-159), and very high (160-200). The Urdu version of the DMSES (U-DMSES) has been validated with moderate to strong psychometric properties (Bijl et al., 1999) (Riaz et al., 2017).
  The U-DMSES will be administered to participants to assess their Self-efficacy in managing Type-II Diabetes, informing interventions to enhance Self-efficacy and overall health and well-being (Luszczynska & Schwarzer, 2015).

CONTACTS AND LOCATIONS:
Locations (1):
- Federal General Hospital, Islamabad, ICT, Pakistan

IPD SHARING:
Plan to Share IPD: No